CLINICAL TRIAL: NCT02001246
Title: An Exploratory Study of Two Intervention Programs for Anger Management for Teens.
Brief Title: Two Anger Management Programs for Teens.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit sufficient numbers of participants to complete the study.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Yoshio Nakamura, Research Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00067796
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Anger; Hostility; Aggression
Keywords: mindfulness; cognitive behavior therapy; awareness; anger; aggression
MeSH Terms: conditions — Aggression | interventions — Anger Management Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Deal program for Anger Management (Active Comparator): The Real Deal Anger Management Program is a structured, video-based intervention, which is an easy-to-implement, "plug and play" program that engages students in: (a) cognitive exercises for learning to recognize and correct thinking errors that lead to anger, (b) active practice of social-behavioral skills through role-playing, and (c) participation in progressive muscle relaxation exercises. The program features three training videos that focus on specific skills for controlling conflict.
  Interventions: Behavioral: Real Deal program for Anger Management
- Mind-body Bridging program (Experimental): The Mind-Body Bridging program for anger management, includes experiential awareness activities, in which individuals learn to become aware of their thoughts, feelings, emotions, and bodily sensations, to help them identify and deal with ruminative and negative thoughts that might be associated with their anger. MBB helps participants use their senses to listen to sounds, and experience visual or tactile input, to calm their minds and relax their bodies. Written 'mapping' exercises enable them to recognize and defuse requirements, which are expectations of how they or the world should be. For the MBB anger management program, participants will be provided with a variety of mapping exercises to identify the source of their anger, and how they can effectively control it.
  Interventions: Behavioral: Mind-body Bridging (MBB) program

INTERVENTIONS:
Behavioral: Real Deal program for Anger Management — Real Deal is an eight week program with sessions one day per week. Each session is approximately 2 hr long.
  Arms: Real Deal program for Anger Management
Behavioral: Mind-body Bridging (MBB) program — MBB is an eight week program with sessions one day per week. Each session is approximately 2 hr long.
  Arms: Mind-body Bridging program

SUMMARY:
The general aim of the proposed pilot study is to evaluate the the efficacy of mind-body bridging (MBB) for anger management compared with the Real Deal anger management program, in helping adolescents control or reduce their anger.

DETAILED DESCRIPTION:
In this pilot randomized-controlled study, we evaluate the effects of MBB as compared with an established anger management program (Real Deal), in helping youth prone to anger develop tools to effectively reduce and control their anger, and potentially reduce other negative emotions and feelings that might be associated with their anger.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* self-, or allo-referred (parents, peers, court-ordered, school, etc.), based on their propensity for displaying various disruptive, externalizing behaviors, including, anger, hostility, oppositional behavior, and temper outbursts, and as such identified by Youth Services (YS) as a suitable candidate to attend a YS anger management program.

Exclusion Criteria:

* none

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Post-assessment in the measure of the Youth Outcomes Questionnaire 30-item (YOQ30) | Baseline (within 1 month of the first session), Mid-assessment (Week 4), Post-Assessment (one week after Week 8)
  The Youth Outcome Questionnaire Self-Report 30 (YOQ-30) is a relatively brief (30-item) psychotherapy outcome measure, which considers general symptoms relevant to many youth mental health disorders and social issues. YOQ-30 is appropriate for tracking youth outcomes over time. It can be completed by adolescents between the ages of 12 and 18 and takes about five minutes to complete. It comprises six subscales (Somatic, Social Isolation, Aggression, Conduct Problems, Hyperactivity/Distractibility, and Depression/ Anxiety). A total score can be computed with 0 indicating no symptomatology and 120 indicating severe symptomatology.
Change from baseline at Post-assessment in the measure of the Brief Aggression Questionnaire (BAQ) | Baseline (within 1 month of the first session), Mid-assessment (Week 4), Post-Assessment (one week after Week 8)
  The BAQ is a 12-item self-report scale identifying four facets of aggression: Physical Aggression, Verbal Aggression, Anger, and Hostility.

SECONDARY OUTCOMES:
Change from baseline at Post-assessment in the measure of Mindfulness | Baseline (within 1 month of the first session), Mid-assessment (Week 4), Post-Assessment (one week after Week 8)
  Five-facet Mindfulness Questionnaire (FFMQ) The FFMQ Short Form (FFMQ-SF) is a 15-item scale assessing five distinct, interpretable facets of mindfulness, including (1) observing, (2) describing, (3) acting with awareness, (4) non-judgement of inner experience, and (5) non-reactivity to inner experience.
Change from baseline at Post-assessment in the measure of Self-compassion | Baseline (within 1 month of the first session), Mid-assessment (Week 4), Post-Assessment (one week after Week 8)
  Self-Compassion Scale (SCS) The SCS short form (SCS-SF) is a 12-item scale used to measure self-compassion, an emotionally positive attitude that can protect against the negative consequences of self-judgment, isolation, and rumination (such as in depression). Self-compassion has three main aspects: (1) self-kindness (being kind and understanding toward oneself in instances of pain or failure, rather than being harshly self-critical); (2) common humanity (perceiving one's experiences as part of the larger human experience, rather than seeing them as separating and isolating); and (3) mindfulness (holding painful thoughts and feelings in balanced awareness, rather than over-identifying with them).

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Nakamura, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Pain Research Center, Anesthesiology, University of Utah, Salt Lake City, Utah
  - Salt Lake County Youth Services, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No